CLINICAL TRIAL: NCT01335607
Title: A Phase I, Open-label Study to Evaluate the Relative Bioavailability of IDX184 and Food Effect in Healthy Male Subjects
Brief Title: A Open-label Study to Evaluate the Relative Bioavailability of Samatasvir (IDX184) and Food Effect in Healthy Male Participants (MK-2355-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2355-006; IDX-08C-006 (Other: Idenix Protocol Number)
Record Dates: First submitted 2011-04-08; First posted 2011-04-14 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — samatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: Samatasvir cap→tab→tab; Part B: cap (Active Comparator): Part A: Samatasvir capsule as a single dose on Day 1 (fasting state) followed by samatasvir tablet as a single dose on Day 8 (fasting state) followed by samatasvir tablet as a single dose on Day 15 (fed state); Part B: samatasvir capsule as a single dose on Day 1 (fed state)
  Interventions: Drug: Samatasvir tablet; Drug: Samatasvir capsule
- Part A: Samatasvir tab→cap→tab; Part B: cap (Active Comparator): Part A: Samatasvir tablet as a single dose on Day 1 (fasting state) followed by samatasvir capsule as a single dose on Day 8 (fasting state) followed by samatasvir tablet as a single dose on Day 15 (fed state); Part B: samatasvir capsule as a single dose on Day 1 (fed state)
  Interventions: Drug: Samatasvir tablet; Drug: Samatasvir capsule

INTERVENTIONS:
Drug: Samatasvir tablet — Two samatasvir (IDX184) 50 mg tablets (100 mg single oral dose)
Drug: Samatasvir capsule — Two samatasvir (IDX184) 50 mg capsules (100 mg single oral dose)

SUMMARY:
The purpose of this study is to:

* Assess the relative bioavailability of 2 oral formulations of samatasvir (capsule and tablet prototype test formulation)
* Compare the amount of study drug that is in the blood after taking either the capsule form of the drug or the tablet form of the drug while fasting.
* Determine the amount of study drug that is in the blood after eating a meal.
* Evaluate the safety of the tablet form of samatasvir in healthy people.

DETAILED DESCRIPTION:
Each participant will receive each of the formulations in a crossover design. Part A Periods 1 and 2: Participants will receive either samatasvir capsules or tablets according to randomization under fasting conditions on Days 1 and 8. Part A Period 3: All participants will receive samatasvir tablets under fed conditons on Day 15.

Each dose will be separated by a 7-day wash-out period. Part B: All participants will receive samatasvir capsules under fed conditons on Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Must be a healthy male with body mass index (BMI) between 18 and 35 kg/m
* Must agree to use an acceptable double-barrier method of birth control.
* Must provide written informed consent after the study has been fully explained.

Exclusion Criteria:

* History of clinically significant diseases, as determined by the investigator.
* Safety laboratory abnormalities at screening which are clinically significant.
* Positive screening test for hepatitis B virus, hepatitis C virus or human immunodeficiency virus (HIV).
* Use of chronic prescription medications within 3 months, acute prescription medications within 14 days, or systemic over-the-counter (OTC) medications within 7 days of the starting the study.
* Current abuse of alcohol or illicit drugs, or history of alcohol or illicit drug abuse within the preceding two years.

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Observed maximum plasma drug concentration (Cmax) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours
Pharmacokinetic parameter: Time to maximum concentration (Tmax) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours
Pharmacokinetic parameter: Area under the drug concentration-time curve from time 0 to last measurable concentration (AUC 0-t) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours
Pharmacokinetic parameter: Area under the drug concentration-time curve from time 0 to 24 hours (AUC 0-24) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours
Pharmacokinetic parameter: Area under the drug concentration-time curve from time 0 to infinity (AUC 0-infinity) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours
Pharmacokinetic parameter: Plasma concentration at 24 hours post dose (C24h) | 24 hours
Pharmacokinetic parameter: Observed plasma terminal half-life (T1/2) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours
Pharmacokinetic parameter: Apparent oral total plasma clearance (CL/F) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours
Pharmacokinetic parameter: Apparent oral total plasma volume of distribution (Vz/F) | Predose (0 hours) and postdose at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours

SECONDARY OUTCOMES:
Percentage of participants who experienced an adverse event | Up to Day 20
Percentage of participants who experienced a serious adverse event | Up to Day 20
Percentage of participants who experienced a Grade 1-4 laboratory abnormality | Up to Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC